CLINICAL TRIAL: NCT04874311
Title: Bintrafusp Alfa and Doxorubicin Hydrochloride in Treating Patients With Advanced Sarcoma. TRUST Study
Brief Title: Bintrafusp Alfa and Doxorubicin Hydrochloride in Treating Patients With Advanced Sarcoma
Acronym: TRUST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB 2020-05; 2020-005703-39 (EudraCT Number)
Record Dates: First submitted 2021-05-04; First posted 2021-05-05 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Advanced Soft-tissue Sarcoma; Metastatic Soft-tissue Sarcoma
Keywords: tertiary lymphoid structure; soft-tissue sarcoma; advanced/metastatic; immunotherapy
MeSH Terms: conditions — Sarcoma; Tertiary Lymphoid Structures; Neoplasm Metastasis | interventions — bintrafusp alfa protein, human; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Arm A: treatment by bintrafusp alfa combined with doxorubicin (Experimental): Soft-tissue sarcoma patients with an inflammed tumor will be treated with bintrafusp alfa combined with doxorubicin for 6 cycles, followed by bintrafusp alfa maintenance
  Interventions: Drug: Bintrafusp alfa; Drug: Doxorubicin
- Standard Arm B: treatment by doxorubicin (Other): Soft-tissue sarcoma patients with an inflammed tumor will be treated with doxorubicin for 6 cycles
  Interventions: Drug: Doxorubicin
- Experimental Arm C: treatment by bintrafusp alfa combined with doxorubicin (Experimental): Soft-tissue sarcoma patients with a cold tumor will be treated with bintrafusp alfa combined with doxorubicin for 6 cycles, followed by bintrafusp alfa maintenance
  Interventions: Drug: Bintrafusp alfa; Drug: Doxorubicin
- Standard Arm D: treatment by doxorubicin (Other): Soft-tissue sarcoma patients with a cold tumor will be treated with doxorubicin for 6 cycles
  Interventions: Drug: Doxorubicin

INTERVENTIONS:
Drug: Bintrafusp alfa — Bintrafusp alfa will be administered by intravenous infusion on day 1 every 3 weeks at a fixed dose of 2400 mg.
  Arms: Experimental Arm A: treatment by bintrafusp alfa combined with doxorubicin; Experimental Arm C: treatment by bintrafusp alfa combined with doxorubicin
Drug: Doxorubicin — Doxorubicin will be administered by intravenous infusion on day 1 every 3 weeks at a fixed dose of 75 mg/m² for a maximum of 6 cycles

SUMMARY:
This study encompasses two multicenter, prospective, open-labeled, 2-arm, non-comparative randomized phase II trials to assess the antitumor activity of bintrafusp alfa in association with doxorubicin

DETAILED DESCRIPTION:
This is a two multicenter, prospective, open-labeled, 2-arm, non-comparative randomized (2:1) phase II trials.

Patients satisfying eligibility criteria will first be stratified into 2 strata / subgroups:

* Soft-tissue sarcoma (STS) patients with an inflamed tumor (i.e. TLS+, defined as presence of mature tertiary lymphoid structures, as per IHC).
* Soft-tissue sarcoma patients with a cold tumor (i.e. TLS-, defined as absence of mature tertiary lymphoid structures, as per IHC).
* Note: TLS+ and TLS- account for 20% and 80% of STS patients, respectively.

STS patients with TLS+ will be randomized between arm A (bintrafusp alfa combined with doxorubicin for 6 cycles, followed by bintrafusp alfa maintenance) and arm B (doxorubicin for 6 cycles) with two patients randomized in arm A for one patient randomized in arm B.

STS patients with TLS- will be randomized between arm C (bintrafusp alfa combined with doxorubicin for 6 cycles, followed by bintrafusp alfa maintenance) and arm D (doxorubicin for 6 cycles) with two patients randomized in arm C for one patient randomized in arm D.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed soft-tissue sarcoma with unknown translocation (including the following histologies but not limited to undifferentiated pleomorphic sarcomas, dedifferentiated liposaromas or leiomyosarcomas). Diagnosis must be reviewed or confirmed by the RRePS Network (Réseau de référence en pathologie des sarcomes et des viscères) as recommended by the French NCI (Institut National du Cancer, Inca).
2. Metastatic or unresectable locally advanced disease,
3. No previous systemic treatment for advanced/metastatic disease,
4. For TLS status: available archived FFPE (Formalin-Fixed Paraffin-Embedded) tumor tissue sample or tumor material newly obtained by biopsy. Except if TLS analysis have been already performed by Biopathological platform at Bergonié Institute, presence or absence of TLS should be confirmed by central review based on FFPE tumor tissue sample (archived or newly obtained by biopsy for research purpose),
5. Age ≥ 18 years,
6. ECOG ≤ 1,
7. Life expectancy > 3 months,
8. Patients must have measurable disease defined as per RECIST v1.1 with at least one lesion that can be measured in at least one dimension as > 10 mm with spiral CT scan.,
9. Patient must comply with the collection of tumor biopsies and biomarkers study. Tumors must be accessible for biopsy,
10. Adequate hematological, renal, metabolic and hepatic function
11. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days prior to randomization. Serum or urine pregnancy test must be repeated within 72 hours prior to receiving the first dose of study medication,
12. Both women and men must agree to use a highly effective method of contraception throughout the treatment period and for at least two months after discontinuation of treatment for women and four months for men.
13. No prior or concurrent malignant disease diagnosed or treated in the last 3 years except for superficial/non-invasive bladder cancer, or basal or squamous cell carcinoma in situ treated with curative intent; b. endoscopically resected GI cancers limited to the mucosal layer without recurrence in > 1 year,
14. Recovery to grade ≤ 1 from any adverse event derived from previous treatment (excluding alopecia and vitiligo of any grade and non-painful peripheral neuropathy grade ≤ 2) according to to NCI-CTCAE, version 5.0,
15. Voluntarily signed and dated written informed consent prior to any study specific procedure,
16. Patients with a social security in compliance with the French law.

Exclusion Criteria:

1. Previous treatment with doxorubicin, daunorubicin, epirubicin, idarubicin and/or any other anthracyclines or anthracediones at the maximum cumulative dose or any approved or investigational treatment targeting PD1, PD-L1 or TGFB1,
2. Known central nervous system malignancy (CNS),
3. Men or women of childbearing potential who are not using an effective method of contraception as previously described; women who are pregnant or breast feeding,
4. Participation to a study involving a medical or therapeutic intervention in the last 30 days,
5. Previous enrolment in the present study,
6. Patient unable to follow and comply with the study procedures because of any geographical, social or psychological reasons,
7. Known hypersensitivity to any involved study drug or any of its formulation components,
8. Any history of anaphylaxis, or recent, within 5 months, history of uncontrollable asthma,
9. Individuals deprived of liberty or placed under legal guardianship,
10. Any of the following cardiac criteria:

    1. Mean resting corrected QT interval (QTcF) ≥ 470 msec, obtained from three consecutive ECGs,
    2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG,
    3. LVEF ≤ 50% per CTCAE v5 by MUGA or echocardiogram
    4. Any factors increasing the risk of QTc prolongation or arrhythmic events such as heart failure, hypokalaemia, potential for torsades de pointes, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years old or any concomitant medication known to prolong the QT interval,
    5. Experience of any of the following procedures or conditions in the preceding 6 months: coronary artery bypass graft, angioplasty, vascular stent, myocardial infarction, unstable angina pectoris, uncontrolled hypertension, congestive heart failure NYHA Grade ≥2, ventricular arrhythmias requiring continuous therapy, supraventricular arrhythmias including atrial fibrillation, which are uncontrolled, haemorrhagic or thrombotic stroke, including transient ischaemic attacks, cerebral vascular accident/stroke or any other central nervous system bleeding
11. Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent:
12. History of bleeding diathesis or recent major bleeding event ,
13. Prior organ transplantation including allogenic stem-cell transplantation, except transplants that do not require immunosuppression,
14. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection requiring systemic therapy, drug-induced interstitial lung disease or subject has had a history of drug-induced pneumonitis that has required oral or IV steroids, and/or other diseases, which in the opinion of the investigator might impair the subject's tolerance for the study or ability to consistently participate in study procedures,
15. Active infection including tuberculosis ,
16. Has known active hepatitis B or hepatitis C,
17. Has a known history of Human Immunodeficiency Virus infection,
18. Receipt of live attenuated vaccine within 30 days prior to the first dose of treatment. Note: Patients, if enrolled, should not receive live vaccine within 30 days prior to the first dose of treatment, whilst receiving study treatments and up to 30 days after the last dose. Seasonal flu vaccines that do not contain a live virus are permitted,
19. Patients with current or history of deep vein thrombosis within 6 months prior to randomization,
20. Any contraindication to biopsy for the research,
21. Any other contraindication to Doxorubicin administration,.
22. Patients with oral anticoagulation therapy based on Vitamin K antagonist.
23. Prior mediastinal radiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Assessment of the antitumor activity of combined administration of standard doxorubicin and double immune modulation with Bintrafusp alfa in terms of 6-month progression-free rate, in STS patients with an inflammed tumor | 6 months
  Antitumor activity will be assessed in terms of 6-month progression-free rate and is defined as the rate of complete or partial response (CR, PR) or stable disease (SD), as per RECIST v1.1.
Assessment of the antitumor activity of combined administration of standard doxorubicin and double immune modulation with Bintrafusp alfa in terms of 6-month progression-free rate, in STS patients with a cold tumor | 6 months
  Antitumor activity will be assessed in terms of 6-month progression-free rate and is defined as the rate of complete or partial response (CR, PR) or stable disease (SD), as per RECIST v1.1.

SECONDARY OUTCOMES:
6-month objective response rate (ORR) independently for patients with an inflammed tumor | 6 months
  Objective response is defined as complete response (CR) or partial response (PR) as per adapted RECIST v1.1.
6-month objective response rate (ORR) independently for patients with a cold tumor | 6 months
  Objective response is defined as complete response (CR) or partial response (PR) as per adapted RECIST v1.1.
Best overall response for patients with an inflammed tumor | throughout the treatment period, an expected average of 6 months
  Best overall response is defined as the best reponse across all time points (RECIST v1.1). The best overall response rate is determined once all the data for the patient is known
Best overall response for patients with a cold tumor | throughout the treatment period, an expected average of 6 months
  Best overall response is defined as the best reponse across all time points (RECIST v1.1). The best overall response rate is determined once all the data for the patient is known
1-year progression-free survival for patients with an inflammed tumor | 1 year
  Progression-free survival is defined as the delay between the date of randomization and the date of progression (as per RECIST v1.1) or death (from any cause), whichever occurs first
1-year progression-free survival for patients with a cold tumor | 1 year
  Progression-free survival is defined as the delay between the date of randomization and the date of progression (as per RECIST v1.1) or death (from any cause), whichever occurs first
1-year overall survival for patients with an inflammed tumor | 1 year
  Overall survival is defined as the delay between the date of randomization and the date of death (from any cause)
1-year overall survival for patients with a cold tumor | 1 year
  Overall survival is defined as the delay between the date of randomization and the date of death (from any cause)
Assessment of the antitumor activity of combined administration of standard doxorubicin and double immune modulation with Bintrafusp alfa in terms of immune response, in STS patients with an inflammed tumor | Throughout the treatment period, an expected average of 6 months
  Immune response is defined following (iRECIST - Seymour et al. 2017).
Assessment of the antitumor activity of combined administration of standard doxorubicin and double immune modulation with Bintrafusp alfa in terms of immune response, in STS patients with a cold tumor | Throughout the treatment period, an expected average of 6 months
  Immune response is defined following (iRECIST - Seymour et al. 2017).
Safety profile independently for each population: Common Terminology Criteria for Adverse Event version 5 | Throughout the treatment period, an expected average of 6 months
  Toxicity graded using the Common Terminology Criteria for Adverse Events version 5

OTHER OUTCOMES:
Tumor immune cells levels independently for each population | baseline, cycle 2 day 1, and progression (each cycle is 21 days)
  Levels of immune cells (CD4, CD8, PDL1)in tumor will be measured by immunohistochemistry
Blood cytokines levels independently for each population | baseline, cycle 2 day 1, cycle 3 day 1 and progression (each cycle is 21 days)
  Levels of cytokines (tryptophane, interleukine) in blood will be measured by ELISA
Blood lymphocytes levels independently for each population | baseline, cycle 2 day 1, cycle 3 day 1 and progression (each cycle is 21 days)
  Levels of fixed PBMC (peripheral blood mononucear cells) in blood will be measured by flow cytometry
Blood kynurenine levels independently for each population | baseline, cycle 2 day 1, cycle 3 day 1 and progression (each cycle is 21 days)
  Levels of kynurenine in blood will be measured by ELISA

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Institut Bergonie, Bordeaux
  - Centre Georges François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmette, Marseille
  - Institut Curie, Paris
  - CHU Poitiers, Poitiers
  - IUCT Oncopole, Toulouse
  - Institut Gustave Roussy, Villejuif